CLINICAL TRIAL: NCT01736163
Title: A Retrospective, Non-interventional Study of Patients With T4 Tumours Comparing the Thyroid Remnant Ablation Success Following Thyrogen and 131I Administration Versus Thyroid Hormone Withdrawal and 131I Administration
Brief Title: A Retrospective Observational Study Comparing Two Different Treatment Options in Thyroid Cancer Patients With T4 Tumours
Status: Completed | Type: Observational
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: THYR04910
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Thyrotropin Alfa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Thyrogen and 131I: Patients were previously treated with Thyrogen in conjunction with a high ablative activity of 131I.
  Interventions: Drug: Thyrogen; Drug: 131I
- Thyroid Hormone Withdrawal and 131I: Patients were previously treated with Thyroid hormone withdrawal (THW) in conjunction with a high ablative activity of 131I.
  Interventions: Drug: 131I; Other: Thyroid Hormone Withdrawal

INTERVENTIONS:
Drug: Thyrogen — 0.9 mg IM, administrated for 2 consecutive days
  Groups: Thyrogen and 131I
Drug: 131I — 28 mCi or ≥ 1.036 GBq.
Other: Thyroid Hormone Withdrawal — Stop taking hormone therapy
  Groups: Thyroid Hormone Withdrawal and 131I

SUMMARY:
The study is to demonstrate non-inferior thyroid remnant first ablation success of Thyrogen and 131I compared to thyroid hormone withdrawal (THW) and 131I in patients with T4 tumour based on historical diagnostic whole body scan (DxWBS) records.

ELIGIBILITY:
Inclusion Criteria:

Historical records from patients who meet all of the following criteria will be eligible for inclusion in this retrospective evaluation:

1. Male or female patients living or deceased, aged 18 years or older at the time of first ablation for thyroid cancer.
2. Diagnosed with a well-differentiated T4 tumour (defined as a primary tumour of any size that extends beyond the thyroid capsule [this may be referred to as TNM classification T4, N0-1, M0-1]). This excludes unusual histological types such as oncocytic (Hurthle cell carcinoma), tall cell, sclerosing or cribriform thyroid cancers.
3. Undergone a near-total or total thyroidectomy on or after 01 January 2000
4. Undergone first ablation of thyroid remnants with high activity 131I (≥28 mCi or ≥ 1.036 GBq).
5. Undergone first 131I ablation for the T4 tumour using either Thyrogen (0.9 mg IM on 2 consecutive days) or THW stimulation. This excludes use of non-standard Thyrogen regimens (i.e., had a regimen of Thyrogen other than the standard 0.9 mg IM on 2 consecutive days or received Thyrogen in combination with THW).
6. Historical records are available confirming ablation results by:

   * DxWBS using small activity (≥2 mCi or 74 MBq) of iodine 131I (or 123I) performed at least 6 months after administration of the first ablation activity of 131I and/or
   * Stimulated Tg measured at least 6 months after administration of the first ablation activity of 131I.

Exclusion Criteria:

Historical records from patients who meet any of the following criteria will be excluded from this retrospective evaluation:

1. Received propylthiouracil, methimazole, vitamins or supplements containing kelp or iodine (taking a multivitamin that does not contain iodine or kelp is acceptable), medications that significantly affect iodine handling such as high dose corticosteroids, high dose diuretics, or lithium in the 45 days before administration of first ablative activity of 131I.
2. Received any iodine-containing contrast agents within 3 months prior to first ablative activity of 131I administered.
3. Used amiodarone within the 2 years prior to first ablative activity of 131I administered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Historical records at clinical sites will be reviewed in a systematic fashion to identify eligible patients.
Sampling Method: Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
First ablation success rate by Diagnostic Whole Body Scan (DxWBS) | at least 6 months after administration of first ablation activity of 131I

SECONDARY OUTCOMES:
First ablation success rate based on stimulated Thyroglobulin (Tg) levels | at least 6 months after administration of first ablation activity of 131I
First ablation success rate based on historical records | at least 6 months after administration of first ablation activity of 131I
Number of adverse events of Thyrogen and 131I arm and THW and 131I arm | Within 30 days of treatment.
  Exploratory safety assessment in patients with T4 tumour for first ablation of thyroid remnants based on historical records.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (9):
- Germany (2):
  - Hanover University School of Medicine, Hanover
  - Klinikum Großhadern, München
- Italy (3):
  - Policlinico S.Orsola-Malpighi, Bologna
  - Instituto Oncologico Veneto, Padua
  - Istituti Fisioterapici Ospitalieri (IFO), Rome
- Portuguese Institute of Oncology, Coimbra, Portugal
- Spain (3):
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Dr Peset, Valencia